CLINICAL TRIAL: NCT01340391
Title: A Wood-plastic Composite Cast - a New Ecological Splinting Method
Brief Title: Safety Study on a Wood-plastic Composite Cast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Nina Lindfors / Senior lecturer, Töölö Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUCS
Record Dates: First submitted 2011-03-28; First posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Distal Radius Fracture
Keywords: cast, radius fracture
MeSH Terms: conditions — Wrist Fractures; Radius Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- splinting method (Experimental): A new splinting method has been invented. This is a study using the splint / cast in treatment of distal radius fractures.
  Interventions: Device: Omnicast

INTERVENTIONS:
Device: Omnicast — dorsal splint 2-5 weeks
  Other Names: Omnicast by Onbone Finland

SUMMARY:
An ecologically friendly and biodegradable wood-plastic composite-cast is studied. Patients, who has sustained a distal radius fracture in need of splinting are requested to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* distal radius fracture not older than 14 days
* age 17-90 years
* mother tongue finnish or swedish

Exclusion Criteria:

* open fracture
* other fractures or a previous fracture
* a previous or simultaneous tendon-, nerve- or vascular injury to the upper extremity
* a multiple injured hand
* decreased co-operation of the patient
* malignancy
* an illness affecting the general health

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
How well will the material fulfil the demands of a splinting material | 1 year
  The aim of the study was to evaluate how well the material fulfils the demands of a splinting material, the subjective satisfaction of the treatment and the orthopaedic technicians´opinion of the material.The following parameters will be detected: immobilisation-time, conservative / operative treatment, re-reposition, mechanical properties of the cast, skin appearance or irritation caused by the cast, allergic reactions and subjective opinion.

CONTACTS AND LOCATIONS:
Overall Officials: Nina C Lindfors, MD, PhD, MSci, Principal Investigator — Helsinki University Central Hospital- Helsinki University